CLINICAL TRIAL: NCT00326170
Title: Phase II Study of the Combination of 5-azacytidine With Valproic Acid and All-trans Retinoic Acid in Patients With High Risk Myelodysplastic Syndrome and Acute Myelogenous Leukemia
Brief Title: Phase II 5-Azacytidine Plus VPA Plus ATRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0799; NCT01575691 (obsolete NCT alias)
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Results first posted 2011-07-11 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Myelodysplastic Syndrome; Acute Myelogenous Leukemia
Keywords: Combination Chemotherapy; MDS; High-Risk Myelodysplastic Syndrome; AML; Acute myelogenous leukemia; valproic acid; VPA; Depakene; 5-azacytidine; 5-aza; Azacitidine; 5-AZC; Vidaza; AZA-CR; Ladakamycin; NSC-102816; All-trans retinoic acid; ATRA; Tretinoin; Vesanoid
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Azacitidine; Valproic Acid; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VPA + 5-aza + ATRA (Experimental): Daily for 7 days, Valproic acid (VPA) starting dose 75 mg/m^2 subcutaneously in combination with 5-azacytidine (5-aza) 50 mg/kg orally; and all-trans retinoic acid (ATRA) 45 mg/m^2 orally daily (in two divided doses) for 5 days starting on day 3.
  Interventions: Drug: 5-Azacytidine (5-aza); Drug: Valproic Acid; Drug: All-Trans Retinoic Acid (ATRA)

INTERVENTIONS:
Drug: 5-Azacytidine (5-aza) — Start at 75 mg/m^2 subcutaneously daily for 7 days.
  Other Names: Azacitidine; 5-azacytidine; 5-AZC; Vidaza; AZA-CR; Ladakamycin; NSC-102816
Drug: Valproic Acid — 50 mg/kg daily by mouth for 7 days, same days as 5-aza.
  Other Names: Depakene
Drug: All-Trans Retinoic Acid (ATRA) — 45 mg/m^2 orally daily (in two divided doses) for 5 days starting on day 3 of the administration of 5-aza and VPA.
  Other Names: Tretinoin (oral); Vesanoid

SUMMARY:
5-aza is a chemotherapy drug with activity in leukemia and myelodysplastic syndromes (MDS). Researchers hope that valproic acid (VPA) and all-trans retinoic acid (ATRA)will increase the effects of 5-aza. The goal of this clinical research study is to find the highest safe dose of valproic acid (VPA) that can be given in combination with 5-azacytidine (5-aza) and all-trans retinoic acid (ATRA) in the treatment of AML and MDS. The safety and effectiveness of this combination therapy will also be studied.

Additional blood and bone marrow samples will be requested. These samples will be used to evaluate the effect of the treatment on leukemic cells. In addition, any leftover blood and bone marrow samples that are collected at the start of the study and during the regularly scheduled evaluations to be sent for research studies. The research studies will examine changes in the blood and bone marrow cells that might help explain the causes of leukemia and MDS and how the combination of 5-aza, VPA, and ATRA works.

DETAILED DESCRIPTION:
Recent studies have shown synergy between demethylating agents and histone deacetylase inhibitors. In my laboratory, we have developed in vitro models using HL-60 and MOLT4 leukemic cells to study the effects of the combination of decitabine (a 5-azacytidine analogue) and valproic acid. Valproic acid is an antiepileptic agent with histone deacetylase inhibitory capacity. These results indicate that the addition of valproic acid to decitabine has an additive effect on growth inhibition, induction of apoptosis, induction of p57KIP2 and p21CIP1 expression independent of cell cycle arrest. These results were dependent on the dose and duration of treatment but not on the sequence used. Based on this data, we developed a phase I/II study of the combination of decitabine and valproic acid (2003-0314) in patients with leukemia that has shown that valproic acid can be safely administered up to doses of 50 mg/kg orally for 10 days in combination with decitabine, and that this combination has significant activity in patients with relapsed/refractory AML and MDS. All-trans retinoic acid (ATRA) is a biological agent that has been shown to induce cell differentiation in leukemia cell lines and has significant clinical activity in acute promyelocytic leukemia with minimal toxicity. In vitro, the combination of ATRA with either a hypomethylating agent or a histone deacetylase inhibitor has been shown to restore ATRA sensitivity in resistant cells. More recently, a German group has reported that the combination of valproic acid and ATRA has activity in patients with MDS and an excellent toxicity profile. 5-azacytidine is a nucleoside analogue with hypomethylating activity that has been shown in a randomized study to benefit patients with MDS, including an improvement in quality of life. Based on this data, this agent was recently approved by the FDA for its use in patients with MDS, and has become the first line agent for patients with MDS that required therapy.

The objectives of the clinical trial are the following:

* To determine the maximal tolerated dose of valproic acid (VPA) in combination with 5-azacytidine (5-aza) and all-trans retinoic acid.
* To determine the clinical activity of the combination of 5-azacytidine, valproic acid and all-trans retinoic acid in patients with AML and MDS.
* To determine the in vivo molecular and biological effects of this combination. These will include analysis of changes in Deoxyribonucleic acid (DNA) methylation, histone modifications, and gene expression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory or relapsed: acute myelogenous leukemia (AML), and myelodysplastic syndrome (MDS) (bone marrow blasts > or = 10%) are eligible.
* Untreated patients older than 60 years of age with AML or MDS (bone marrow blasts > or = 10%) who refuse or are not eligible for front-line chemotherapy, are eligible.
* Performance status of < or = 2 by the Eastern Cooperative Oncology Group (ECOG) scale.
* Signed informed consent indicating that patients are aware of the investigational nature of this study in keeping with the policies of University of Texas M D Anderson Cancer Center (UTMDACC).
* Age > 2 years. Valproic acid has been associated with a higher rate of severe liver toxicity in children younger than 2 years.
* Patients must have been off chemotherapy for 2 weeks prior to entering this study and recovered from the toxic effects of that therapy, unless there is evidence of rapidly progressive disease. Use of hydroxyurea for patients with rapidly proliferative disease is allowed for the first two weeks on therapy.
* Adequate liver function (bilirubin of < 2mg/dL, SGPT < 3 * ULN) and renal function (creatinine < 2mg/dL).
* Women of childbearing potential must practice contraception. Men and women must continue birth control for the duration of the trial.
* Patients with relapsed /refractory disease with inv16, t(8;21) or t(15;17) are eligible.

Exclusion Criteria:

* Nursing and pregnant females are excluded.
* Patients with active and uncontrolled infections are excluded.
* Patients already receiving valproic acid or receiving other anticonvulsants will be excluded.
* Untreated patients younger than 60 years will not be candidates for this study.
* Patients with untreated disease inv16, t(8;21) or t(15;17) will be excluded.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-07; Primary Completion 2007-07 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Soriano AO, Yang H, Faderl S, Estrov Z, Giles F, Ravandi F, Cortes J, Wierda WG, Ouzounian S, Quezada A, Pierce S, Estey EH, Issa JP, Kantarjian HM, Garcia-Manero G. Safety and clinical activity of the combination of 5-azacytidine, valproic acid, and all-trans retinoic acid in acute myeloid leukemia and myelodysplastic syndrome. Blood. 2007 Oct 1;110(7):2302-8. doi: 10.1182/blood-2007-03-078576. Epub 2007 Jun 27. PMID 17596541
- See also: M.D. Anderson's internet website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 06/10/05 through 11/17/06. All participants recruited at UT MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | VPA + 5-aza + ATRA
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | VPA + 5-aza + ATRA
Number analyzed (Participants) | 34
Age Continuous [Median (Full Range); unit: years] | 70 [49 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response
Description: Clinical activity of combination defined as: Complete Response (CR), bone marrow with 5% or fewer blasts and peripheral blood count with an absolute neutrophil count of 10^9/L or more and platelet count of 100x10^9 or more; Complete response without platelets (CRp), a complete response except for a platelet count less than 100x10^9 and transfusion independent; and Bone Marrow (BM) Response, bone marrow blast of 5% or less but without meeting the peripheral blood count criteria for (CR) or (CRp).
Time Frame: Up to 12 cycles of treatment (28 day cycles)
Measure: Number; unit: Participants
Arm/Group | VPA + 5-aza + ATRA
Number analyzed (Participants) | 34
Participants
  CR | 12
  CRp | 3
  BM | 7

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | VPA + 5-aza + ATRA
Serious Adverse Events (participants affected / at risk) | 31/34
Other Adverse Events (participants affected / at risk) | 11/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VPA + 5-aza + ATRA (N=34)
Infection (Infections and infestations) | 8 (8)
Death (General disorders) | 11 (11)
Fatigue (General disorders) | 7 (8)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Somnolence (Nervous system disorders) | 10 (11)
Syncope (Nervous system disorders) | 2 (2)
Confusion (Nervous system disorders) | 4 (4)
Pain (General disorders) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Dehydration (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Hemorrhage (Vascular disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Edema (Blood and lymphatic system disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VPA + 5-aza + ATRA (N=34)
Weakness (General disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Confusion (Nervous system disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes